CLINICAL TRIAL: NCT00855465
Title: Randomized, Double-blind, Placebo-controlled, Multi-centre, Multi-national Study to Evaluate the Efficacy and Safety of Oral BAY63-2521 (1 mg, 1.5 mg, 2 mg, or 2.5 mg Tid) in Patients With Chronic Thromboembolic Pulmonary Hypertension (CTEPH)
Brief Title: A Study to Evaluate Efficacy and Safety of Oral BAY63-2521 in Patients With CTEPH.
Acronym: CHEST-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11348; 2007-000072-16 (EudraCT Number)
Record Dates: First submitted 2008-12-15; First posted 2009-03-04 (Estimated); Results first posted 2014-03-11 (Estimated); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Hypertension
Keywords: Chronic thromboembolic pulmonary hypertension; PH; soluble Guanylate Cyclase Stimulator; sGC
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — riociguat

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Riociguat (Adempas, BAY63-2521)_individual dose titration (Experimental): Participants received Riociguat orally as a film-coated tablet up to 2.5mg three times daily (tid) (titration between 1.0 mg and 2.5 mg tid based on an individual dose titration (IDT) scheme) for 16 weeks
  Interventions: Drug: Riociguat (Adempas, BAY63-2521)
- Placebo (Placebo Comparator): Participants received Placebo orally as a film-coated tablet three times daily (tid) for 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Riociguat (Adempas, BAY63-2521) — BAY63-2521: 1 mg tid - 2,5 mg tid orally for 16 weeks.
  Arms: Riociguat (Adempas, BAY63-2521)_individual dose titration
Drug: Placebo — Matching Placebo tid orally for 16 weeks
  Arms: Placebo

SUMMARY:
The aim of the study is to assess the efficacy and safety of different doses of BAY63-2521, given orally for 16 weeks, in patients with Chronic Thromboembolic Pulmonary Hypertension (CTEPH).

DETAILED DESCRIPTION:
Adverse event data will be covered in Adverse events section.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with CTEPH either inoperable or with persistent or recurrent PH after surgery.

Exclusion Criteria:

* All types of pulmonary hypertension except subtypes 4.1 and 4.2 of the Venice Clinical Classification of Pulmonary Hypertension.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2009-02-23 (Actual); Primary Completion 2012-06-27 (Actual); Study Completion 2012-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (83):
- United States (9):
  - La Jolla, California
  - Sacramento, California
  - Miami, Florida
  - Iowa City, Iowa
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dallas, Texas
- Corrientes, Argentina
- Prahran, Victoria, Australia
- Austria (2):
  - Innsbruck
  - Vienna
- Belgium (2):
  - Bruxelles - Brussel
  - Leuven
- Brazil (3):
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo
  - Rio de Janeiro
- Canada (5):
  - Calgary, Alberta
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- China (3):
  - Qingdao, Shandong
  - Beijing
  - Shanghai
- Vseobecna fakultni nemocnice, Prague, Czechia
- Aarhus N, Denmark
- France (8):
  - Brest
  - Caen
  - Hopital Antoine Beclere, Clamart
  - Lille
  - Nice
  - Pessac
  - Rouen
  - Vandœuvre-lès-Nancy
- Germany (11):
  - Heidelberg, Baden-Wurttemberg
  - München, Bavaria
  - Würzburg, Bavaria
  - Giessen, Hesse
  - Hanover, Lower Saxony
  - Greifswald, Mecklenburg-Vorpommern
  - Cologne, North Rhine-Westphalia
  - Homburg, Saarland
  - Dresden, Saxony
  - Leipzig, Saxony
  - Hamburg
- Pavia, Lombardy, Italy
- Japan (14):
  - Nagoya, Aichi-ken
  - Seto, Aichi-ken
  - Kitakyushu, Fukuoka
  - Komatsu, Ishikawa-ken
  - Fujisawa, Kanagawa
  - Kawasaki, Kanagawa
  - Sendai, Miyagi
  - Suwa, Nagano
  - Suita, Osaka
  - Bunkyo-ku, Tokyo
  - Mitaka, Tokyo
  - Shinjuku-ku, Tokyo
  - Chiba
  - Fukuoka
- Mexico (3):
  - Monterrey, Nuevo León
  - Mexico City
  - Querétaro
- Amsterdam, Netherlands
- Poland (2):
  - Krakow
  - Otwock
- Coimbra, Portugal
- Russia (2):
  - Novosibirsk
  - Saint Petersburg
- Bratislava, Slovakia
- Seoul, South Korea
- Spain (2):
  - Barcelona
  - Madrid
- Zurich, Switzerland
- Taipei, Taiwan
- Turkey (Türkiye) (3):
  - Ankara
  - Istanbul
  - Izmir
- United Kingdom (3):
  - Cambridge, Cambridgeshire
  - Glasgow, West Dunbartonshire
  - London

REFERENCES:
- [Result] Ghofrani HA, D'Armini AM, Grimminger F, Hoeper MM, Jansa P, Kim NH, Mayer E, Simonneau G, Wilkins MR, Fritsch A, Neuser D, Weimann G, Wang C; CHEST-1 Study Group. Riociguat for the treatment of chronic thromboembolic pulmonary hypertension. N Engl J Med. 2013 Jul 25;369(4):319-29. doi: 10.1056/NEJMoa1209657. PMID 23883377
- [Result] Archer SL. Riociguat for pulmonary hypertension--a glass half full. N Engl J Med. 2013 Jul 25;369(4):386-8. doi: 10.1056/NEJMe1306684. No abstract available. PMID 23883383
- [Result] Simonneau G, D'Armini AM, Ghofrani HA, Grimminger F, Jansa P, Kim NH, Mayer E, Pulido T, Wang C, Colorado P, Fritsch A, Meier C, Nikkho S, Hoeper MM. Predictors of long-term outcomes in patients treated with riociguat for chronic thromboembolic pulmonary hypertension: data from the CHEST-2 open-label, randomised, long-term extension trial. Lancet Respir Med. 2016 May;4(5):372-80. doi: 10.1016/S2213-2600(16)30022-4. Epub 2016 Apr 8. PMID 27067478
- [Result] Wang C, Jing ZC, Huang YG, Zhou DX, Liu ZH, Meier C, Nikkho S, Curram J, Zhang P, He JG. Riociguat for the treatment of pulmonary hypertension: Chinese subgroup analyses and comparison. Heart Asia. 2016 May 17;8(1):74-82. doi: 10.1136/heartasia-2015-010712. eCollection 2016. PMID 27326239
- [Result] Ghofrani HA, Humbert M, Langleben D, Schermuly R, Stasch JP, Wilkins MR, Klinger JR. Riociguat: Mode of Action and Clinical Development in Pulmonary Hypertension. Chest. 2017 Feb;151(2):468-480. doi: 10.1016/j.chest.2016.05.024. Epub 2016 Jun 2. PMID 27263466
- [Result] Kim DY, Kim HJ, Han KH, Han SY, Heo J, Woo HY, Um SH, Kim YH, Kweon YO, Lim HY, Yoon JH, Lee WS, Lee BS, Lee HC, Ryoo BY, Yoon SK. Real-Life Experience of Sorafenib Treatment for Hepatocellular Carcinoma in Korea: From GIDEON Data. Cancer Res Treat. 2016 Oct;48(4):1243-1252. doi: 10.4143/crt.2015.278. Epub 2016 Feb 24. PMID 26910470
- [Result] Kudo M, Ikeda M, Takayama T, Numata K, Izumi N, Furuse J, Okusaka T, Kadoya M, Yamashita S, Ito Y, Kokudo N. Safety and efficacy of sorafenib in Japanese patients with hepatocellular carcinoma in clinical practice: a subgroup analysis of GIDEON. J Gastroenterol. 2016 Dec;51(12):1150-1160. doi: 10.1007/s00535-016-1204-2. Epub 2016 Apr 22. PMID 27106231
- [Result] Benza RL, Boucly A, Farber HW, Frost AE, Ghofrani HA, Hoeper MM, Lambelet M, Rahner C, Bansilal S, Nikkho S, Meier C, Sitbon O. Change in REVEAL Lite 2 risk score predicts outcomes in patients with pulmonary arterial hypertension in the PATENT study. J Heart Lung Transplant. 2022 Mar;41(3):411-420. doi: 10.1016/j.healun.2021.10.013. Epub 2021 Oct 28. PMID 34848133
- [Result] Benza RL, Farber HW, Frost AE, Ghofrani HA, Corris PA, Lambelet M, Nikkho S, Meier C, Hoeper MM. Application of the REVEAL risk score calculator 2.0 in the CHEST study. Respir Med. 2022 Apr-May;195:106783. doi: 10.1016/j.rmed.2022.106783. Epub 2022 Mar 1. PMID 35256218
- [Derived] Kim NH, D'Armini AM, Grimminger F, Grunig E, Hoeper MM, Jansa P, Mayer E, Neurohr C, Simonneau G, Torbicki A, Wang C, Fritsch A, Davie N, Ghofrani HA. Haemodynamic effects of riociguat in inoperable/recurrent chronic thromboembolic pulmonary hypertension. Heart. 2017 Apr;103(8):599-606. doi: 10.1136/heartjnl-2016-309621. Epub 2016 Dec 23. PMID 28011757
- [Derived] Saleh S, Becker C, Frey R, Muck W. Population pharmacokinetics and the pharmacokinetic/pharmacodynamic relationship of riociguat in patients with pulmonary arterial hypertension or chronic thromboembolic pulmonary hypertension. Pulm Circ. 2016 Mar;6(Suppl 1):S86-96. doi: 10.1086/685404. PMID 27162632

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only subjects with symptomatic chronic thromboembolic pulmonary hypertension (CTEPH) could participate in this study. CTEPH was defined either as inoperable or as persisting or recurrent PH after pulmonary endarterectomy.
Pre-assignment Details: 446 subjects were screened in 89 study centers in 26 countries worldwide. 184 of the 446 screened subjects were not randomized (adverse event [1], death [4], protocol violation [164], withdrawal by subject [15]). 262 of the 446 subjects were randomized. 261 of the 262 randomized subjects received study medication.
Period: Treatment Period
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Started | 174 | 88
Participants Received Treatment | 173 (1 subject randomized but not treated) | 88
Completed | 160 | 83
Not Completed | 14 | 5
Not completed — Adverse Event | 4 | 2
Not completed — Death | 2 | 2
Not completed — Lack of Efficacy | 2 | 1
Not completed — Non-compliance | 1 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Not treated | 1 | 0
Period: Follow-up Period (FUP)
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Started | 17 (Started FUP only if prematurely withdrawn from trt period or if not entering LTE study.) | 4 (Started FUP only if prematurely withdrawn from trt period or if not entering LTE study.)
Completed | 9 | 2
Not Completed | 8 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Missing | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo | Total
Number analyzed (Participants) | 173 | 88 | 261
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.3 (13.9) | 59.2 (12.7) | 59.3 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 54 | 172
  Male | 55 | 34 | 89
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 120 | 65 | 185
  Black or African American | 7 | 1 | 8
  Asian | 37 | 20 | 57
  Mixed | 1 | 0 | 1
  Not reported | 8 | 2 | 10
Operability [Number; unit: Participants] — CTEPH defined as inoperable or as persisting/recurrent PH after pulmonary endarterectomy (PEA).
  Participants
    Inoperable CTEPH | 121 | 68 | 189
    Postoperative CTEPH | 52 | 20 | 72
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.13 (5.75) | 27.73 (5.30) | 27.33 (5.60)
6-minute walking distance [Mean (Standard Deviation); unit: Meters] — 6-minute walking distance (6MWD) is a measure for the objective evaluation of a participant's functional exercise capacity.
  Meters | 342.3 (81.9) | 356.0 (74.7) | 346.9 (79.7)
WHO (World Health Organization) functional class [Number; unit: Participants] — The WHO functional assessment of pulmonary arterial hypertension ranged from functional class I (Patients with PH but without resulting limitation of physical activity) to class IV (Patients with PH with inability to carry out any physical activity without symptoms. These patients manifest signs of right-heart failure.). Changes to a lower WHO functional class resemble improvement; changes to a higher functional class resemble deterioration of pulmonary arterial hypertension (PAH).
  Participants
    missing | 0 | 1 | 1
    I | 3 | 0 | 3
    II | 55 | 25 | 80
    III | 107 | 60 | 167
    IV | 8 | 2 | 10
Pulmonary vascular resistance [Mean (Standard Deviation); unit: dyn*s*cm^-5] — The pulmonary vascular resistance (PVR) is a calculated hemodynamic parameter. PVR is derived from the directly measured parameters mean pulmonary arterial pressure (PAPmean) and pulmonary capillary wedge pressure (PCWP), divided by the cardiac output (CO). PVR and PAPmean are acquired during a right heart catheterization. CO is a calculated hemodynamic parameter, too. Formula: PVR = 80*(PAPmean - PCWP)/CO
  dyn*s*cm^-5 | 790.68 (431.57) | 779.32 (400.94) | 786.68 (420.21)

OUTCOME MEASURES:

1. Primary Outcome: 6 Minutes Walking Distance (6MWD) - Change From Baseline to Week 16
Description: 6-minute walking distance (6MWD) is a measure for the objective evaluation of a participant's functional exercise capacity.
Time Frame: Baseline and week 16
Population: Intent to Treat (ITT) - a randomized participant was valid for ITT analyses if at least one dose of study medication was administered.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 173 | 88
Meters | 38.9 (79.3) | -5.5 (84.3)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521)_individual Dose Titration vs Placebo; Missing values for participants who withdrew/died before 16 weeks were imputed with a worst value of 0m in case of death/clinical worsening without termination visit and with the last observed value otherwise. Comparison was done using analysis of covariance (ANCOVA), with baseline 6MWD as a covariate and treatment group and region as main effects. The primary statistical method was the stratified Wilcoxon test if the Shapiro-Wilk test for normality of residuals was statistically significant; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — Prespecified significance level for all significance tests was 5%. Primary analysis, due to result of Shapiro-Wilk test; Test was stratified by region
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521)_individual Dose Titration vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — Additional analysis, due to result of Shapiro-Wilk test; Mean Difference (Final Values) = 45.69, 95% CI 2-sided [24.74 to 66.63]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521)_individual Dose Titration vs Placebo; Shapiro-Wilk test for normality of ANCOVA residuals; Test type: Superiority or Other; p = 0.0001, Shapiro-Wilk

2. Secondary Outcome: Pulmonary Vascular Resistance (PVR) - Change From Baseline to Week 16
Description: The pulmonary vascular resistance (PVR) is a calculated hemodynamic parameter. PVR is derived from the directly measured parameters mean pulmonary arterial pressure (PAPmean) and pulmonary capillary wedge pressure (PCWP), divided by the cardiac output (CO). PVR and PAPmean are acquired during a right heart catheterization. CO is a calculated hemodynamic parameter, too. Formula: PVR = 80*(PAPmean - PCWP)/CO
Time Frame: Baseline and week 16
Population: Intent to Treat (ITT) - a randomized participant was valid for ITT analyses if at least one dose of study medication was administered. Only participants with a baseline and at least one post-baseline measurement were included in the analysis of PVR.
Measure: Mean (Standard Deviation); unit: dyn*s*cm^-5
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 151 | 82
dyn*s*cm^-5 | -225.68 (247.52) | 23.07 (273.53)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521)_individual Dose Titration vs Placebo; Missing values at week 16 were imputed using the last available post-baseline observation. Same analysis method as for primary efficacy parameter; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — Hierarchical testing for secondary efficacy parameters in the order: PVR, NT-proBNP, WHO functional class, Time to clinical worsening, Borg scale, EQ5D, LPH. Primary analysis due to result of Shapiro-Wilk test
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521)_individual Dose Titration vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — Additional analysis due to result of Shapiro-Wilk test; Mean Difference (Final Values) = -246.43, 95% CI 2-sided [-303.33 to -189.53]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521)_individual Dose Titration vs Placebo; Shapiro-Wilk test for normality of ANCOVA residuals; Test type: Superiority or Other; p = 0.0001, Shapiro-Wilk

3. Secondary Outcome: N-terminal Prohormone of Brain Natriuretic Peptide (NT-proBNP) - Change From Baseline to Week 16
Description: N-terminal pro-brain natriuretic peptide (NT-proBNP) levels in the blood are used for screening, diagnosis of acute congestive heart failure (CHF) and may be useful to establish prognosis in heart failure.
Time Frame: Baseline and week 16
Population: Intent to Treat (ITT) - a randomized participant was valid for ITT analyses if at least one dose of study medication was administered. Only participants with a baseline and at least one post-baseline measurement were included in the analysis of NT-proBNP.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 150 | 73
pg/mL | -290.69 (1716.90) | 76.35 (1446.63)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521)_individual Dose Titration vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521)_individual Dose Titration vs Placebo; Test type: Superiority or Other; p = 0.0293, ANCOVA — Additional analysis due to result of Shapiro-Wilk test; Mean Difference (Final Values) = -443.99, 95% CI 2-sided [-842.95 to -45.03]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521)_individual Dose Titration vs Placebo; Shapiro-Wilk test for normality of ANCOVA residuals; Test type: Superiority or Other; p = 0.0001, Shapiro-Wilk

4. Secondary Outcome: World Health Organization (WHO) Functional Class - Change From Baseline to Week 16
Description: The WHO functional assessment of pulmonary arterial hypertension ranged from functional class I (Patients with PH but without resulting limitation of physical activity) to class IV (Patients with PH with inability to carry out any physical activity without symptoms. These patients manifest signs of right-heart failure.). Changes to a lower WHO functional class resemble improvement; changes to a higher functional class resemble deterioration of PAH.
Time Frame: Baseline and week 16
Population: Intent to Treat (ITT) - a randomized participant was valid for ITT analyses if at least one dose of study medication was administered. Participants with a missing baseline were excluded from the analysis of WHO functional class.
Measure: Number; unit: Percentage of Participants
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 173 | 87
Percentage of Participants
  -2 | 2.3 | 0
  -1 | 30.6 | 14.9
  0 | 61.8 | 78.2
  1 | 4.0 | 3.4
  2 | 0.6 | 3.4
  3 | 0.6 | 0
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521)_individual Dose Titration vs Placebo; Missing values for participants who withdrew or died before 16 weeks were imputed with a worst value of IV in case of clinical worsening without termination visit or measurement at that termination visit and with a worst value of V in case of death and with the last observed value otherwise; Test type: Superiority or Other; p = 0.0026, Wilcoxon (Mann-Whitney) — Hierarchical testing for secondary efficacy parameters in the order: PVR, NT-proBNP, WHO functional class, Time to clinical worsening, Borg scale, EQ5D, LPH; Test was stratified by region

5. Secondary Outcome: Percentage of Participants With Clinical Worsening
Description: The combined endpoint "time to clinical worsening", made up of the following components, defined by the first occurrence: all-cause mortality; heart/lung transplantation; rescue endarterectomy; first hospitalization due to pulmonary hypertension; start of a new pulmonary hypertension treatment; persistent worsening of 6MWD or WHO functional class due to deterioration of PH.
Time Frame: At week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 173 | 88
Percentage of participants
  Any Event | 2.3 | 5.7
  Hospitalization due to pulmonary hypertension | 0 | 1.1
  Start of new pulmonary hypertension | 1.2 | 1.1
  Decrease in 6MWT due to pulmonary hypertension | 0.6 | 2.3
  Persistant worsening of functional class due to PH | 0 | 1.1
  Death | 1.2 | 3.4
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521)_individual Dose Titration vs Placebo; Test for difference of occurence of "Any event"; Test type: Superiority or Other; p = 0.1724, Log Rank — [p-value comment as in outcome 4, analysis 1]; Test was stratified by region; Risk Difference (RD) = -3.37, 95% CI 2-sided [-8.72 to 1.99] — Based on Mantel-Haenszel estimate stratified by region

6. Secondary Outcome: Borg CR 10 Scale - Change From Baseline to Week 16
Description: The Borg CR10 Scale is a participant reported outcome measure used in clinical diagnosis of e.g. breathlessness and dyspnea. It documents the participant's exertion during a physical test. Low values indicate low levels of exertion; high values indicate more intense exertion reported by the participant. The score ranges from 0 ("Nothing at all") to 10 ("Extremely strong - Maximal").
Time Frame: Baseline and week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 173 | 88
Scores on a scale | -0.83 (2.39) | 0.17 (2.42)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521)_individual Dose Titration vs Placebo; Missing values for participants who withdrew or died before 16 weeks were imputed with a worst value of 10 in case of death or clinical worsening without termination visit and with the last observed value otherwise; Test type: Superiority or Other; p = 0.0035, Wilcoxon (Mann-Whitney) — Hierarchical testing for secondary efficacy parameters in the order: PVR, NT-proBNP, WHO functional class, Time to clinical worsening, Borg scale, EQ5D, LPH. Nominally significant only due to hierarchical testing; Test was stratified by region

7. Secondary Outcome: EQ-5D Utility Score - Change From Baseline to Week 16
Description: EQ-5D utility score is a Quality-of-Life participant reported outcome measure. The utility score is calculated based on five questions concerning problems with mobility, self-care, usual activities, pain/discomfort and anxiety/depression. An increase in the utility score represents an improvement in quality of life. The score ranges from -0.594 (worst answer in all five questions) to 1 (best answer in all five questions).
Time Frame: Baseline and week 16
Population: Intent to Treat (ITT) - a randomized participant was valid for ITT analyses if at least one dose of study medication was administered. Participants with a missing baseline were excluded from the analysis of the EQ5D utility score.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 172 | 87
Scores on a scale | 0.0615 (0.2768) | -0.0819 (0.3446)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521)_individual Dose Titration vs Placebo; Missing values at baseline were imputed using last available observation prior to start of study treatment. Missing values for participants who withdrew or died before 16 weeks were imputed with a worst value of -0.594 in case of death or clinical worsening without termination visit and with the last observed value otherwise; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — Hierarchical testing for secondary efficacy parameters in the order: PVR, NT-proBNP, WHO FC, TTCW, Borg scale, EQ5D, LPH. Primary analysis due to result of Shapiro-Wilk test.Nominally significant only due to hierarchical testing
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521)_individual Dose Titration vs Placebo; Test type: Superiority or Other; p = 0.0002, ANCOVA — Additional analysis due to result of Shapiro-Wilk test; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [0.06 to 0.21]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521)_individual Dose Titration vs Placebo; Shapiro-Wilk test for normality of ANCOVA residuals; Test type: Superiority or Other; p = 0.0001, Shapiro-Wilk

8. Secondary Outcome: Living With Pulmonary Hypertension (LPH) Questionnaire - Change From Baseline to Week 16
Description: The self-reported Living with Pulmonary Hypertension (LPH) questionnaire is designed to measure the effects of PH and PH-specific treatments on an individual's quality of life. The LPH total score can range from 0 (best) to 105 (worst).
Time Frame: Baseline and week 16
Population: Intent to Treat (ITT) - a randomized participant was valid for ITT analyses if at least one dose of study medication was administered. Participants with a missing baseline were excluded from the analysis of the LPH questionnaire.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 170 | 86
Scores on a scale | -6.72 (18.62) | -2.09 (19.31)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521)_individual Dose Titration vs Placebo; Missing values at baseline were imputed using last available observation prior to start of study treatment. Missing values for participants who withdrew or died before 16 weeks were imputed with a worst value of 105 in case of death or clinical worsening without termination visit and with the last observed value otherwise; Test type: Superiority or Other; p = 0.1220, Wilcoxon (Mann-Whitney) — Hierarchical testing for secondary efficacy parameters in the order: PVR, NT-proBNP, WHO functional class, Time to clinical worsening, Borg Dyspnea Score, EQ5D, LPH. Primary analysis due to result of Shapiro-Wilk test
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521)_individual Dose Titration vs Placebo; Test type: Superiority or Other; p = 0.0165, ANCOVA — Additional analysis due to result of Shapiro-Wilk test; Mean Difference (Final Values) = -5.76, 95% CI 2-sided [-10.45 to -1.06]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521)_individual Dose Titration vs Placebo; Shapiro-Wilk test for normality of ANCOVA residuals; Test type: Superiority or Other; p = 0.0001, Shapiro-Wilk

9. Other Pre Specified Outcome: All Caused Mortality
Description: All cause mortality (including cardiovascular mortality) was one component of the composite endpoint "time to clinical worsening".
Time Frame: At visit 6 (week 16)
Population: Intent to Treat (ITT) - a randomized subject was valid for ITT analyses if at least one dose of study medication was administered.
Measure: Number; unit: Participants
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 173 | 88
Participants | 2 | 3

10. Other Pre Specified Outcome: Mean Pulmonary Artery Pressure (PAPmean) - Change From Baseline to Week 16
Description: Mean pulmonary arterial pressure (PAPmean) is a directly measured hemodynamic parameter. PAPmean is recorded during a right heart catheterization.
Time Frame: Baseline and week 16
Population: Intent to Treat (ITT) - a randomized participant was valid for ITT analyses if at least one dose of study medication was administered.
  Only participants with a baseline and at least one post-baseline measurement were included in the analysis of PAPmean.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 156 | 84
mmHg | -4.31 (6.70) | 0.76 (7.26)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521)_individual Dose Titration vs Placebo; Missing values at week 16 were imputed using the last available post-baseline observation. Same analysis as for primary efficacy parameter; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — Exploratory testing. Primary analysis due to result of Shapiro-Wilk test
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521)_individual Dose Titration vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — Additional analysis due to result of Shapiro-Wilk test; Mean Difference (Final Values) = -4.96, 95% CI 2-sided [-6.75 to -3.16]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521)_individual Dose Titration vs Placebo; Shapiro-Wilk test for normality of ANCOVA residuals; Test type: Superiority or Other; p = 0.0231, Shapiro-Wilk

11. Other Pre Specified Outcome: Cardiac Index (CI) - Change From Baseline to Week 16
Description: The cardiac index (CI) is a calculated hemodynamic parameter. CI is derived from the directly measured parameters cardiac output (CO), divided by the body surface area (BSA). BSA is a calculated parameter, using the subject's height and weight in the DuBois formula. Formula: BSA = (W [kg]*0.425)*(H [cm]*0.725)*0.007184 (m^2)
Time Frame: Baseline and week 16
Population: Intent to Treat (ITT) - a randomized participant was valid for ITT analyses if at least one dose of study medication was administered.
  Only participants with a baseline and at least one post-baseline measurement were included in the analysis of CI.
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 155 | 83
L/min/m^2 | 0.45 (0.56) | -0.01 (0.58)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521)_individual Dose Titration vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Exploratory testing. Primary analysis due to result of Shapiro-Wilk test; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [0.33 to 0.62]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521)_individual Dose Titration vs Placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — Additional analysis due to result of Shapiro-Wilk test
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521)_individual Dose Titration vs Placebo; Shapiro-Wilk test for normality of ANCOVA residuals; Test type: Superiority or Other; p = 0.1160, Shapiro-Wilk

12. Other Pre Specified Outcome: Systolic Blood Pressure (SBP) - Change From Baseline to Week 16
Description: Systolic systemic arterial blood pressure (SBP) is a directly non-invasively measured hemodynamic parameter. Range allowed in this study at Visit 0 and/or Visit 1 before randomization: 95 - 180 mmHg.
Time Frame: Baseline and week 16
Population: Safety (SAF) - a randomized participant was valid for safety analyses if at least one dose of study medication was administered.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 173 | 88
mmHg | -10.49 (14.17) | -5.28 (14.61)

13. Other Pre Specified Outcome: Diastolic Blood Pressure (DBP) - Change From Baseline to Week 16
Description: Diastolic systemic arterial blood pressure (DBP) is a directly non-invasively measured hemodynamic parameter. Range allowed in this study at Visit 0 and/or Visit 1 before randomization: <= 110 mmHg.
Time Frame: Baseline and week 16
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 173 | 88
mmHg | -8.17 (10.81) | -3.40 (10.38)

14. Other Pre Specified Outcome: Heart Rate (HR) - Change From Baseline to Week 16
Description: Heart rate (HR) is a directly non-invasively measured hemodynamic parameter. Range allowed in this study at Visit 0 and/or Visit 1 before randomization: 50 -105 beats per minute (bpm) at rest.
Time Frame: Baseline and week 16
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Beats/min
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 173 | 88
Beats/min | 0.83 (11.74) | 1.67 (12.37)

15. Other Pre Specified Outcome: Alanine Aminotransferase (ALT) - Change From Baseline to Week 16
Description: Alanine Aminotransferase (ALT) is a standard clinical chemistry parameter. Normal range: 0 to 45 U/L.
Time Frame: Baseline and week 16
Population: Safety (SAF) - a randomized participant was valid for safety analyses if at least one dose of study medication was administered. Only participants with a baseline and at least one measurement on treatment (or up to two days after stopping treatment) were included in the analysis of laboratory parameters.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 161 | 82
U/L | -1.2 (16.2) | 2.2 (13.6)

16. Other Pre Specified Outcome: Aspartate Aminotransferase (AST) - Change From Baseline to Week 16
Description: Aspartate Aminotransferase (AST) is a standard clinical chemistry parameter. Normal range: 0 to 41 U/L.
Time Frame: Baseline and week 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 160 | 82
U/L | 0.3 (14.4) | 2.8 (12.0)

17. Other Pre Specified Outcome: Alkaline Phosphatase (AP) - Change From Baseline to Week 16
Description: Alkaline phosphatase (AP) is a standard clinical chemistry parameter. Normal range: 40 to 129 U/L (males), 35 to 104 U/L (females)
Time Frame: Baseline and week 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 162 | 82
U/L | -3.8 (19.4) | 2.5 (20.2)

18. Other Pre Specified Outcome: Bilirubin - Change From Baseline to Week 16
Description: Bilirubin is a standard clinical chemistry parameter. Normal range: 0.1 to 1.2 mg/dL
Time Frame: Baseline and week 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 162 | 82
mg/dL | 0.010 (0.483) | 0.189 (0.453)

19. Other Pre Specified Outcome: Creatinine - Change From Baseline to Week 16
Description: Creatinine is a standard clinical chemistry parameter. Normal range: 0.25 to 1.20 mg/dL (males), 0.46 to 1.00 mg/dL (females)
Time Frame: Baseline and week 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 162 | 82
mg/dL | 0.003 (0.338) | 0.032 (0.178)

20. Other Pre Specified Outcome: Creatinine Clearance - Change From Baseline to Week 16
Description: Creatinine clearance is a standard clinical chemistry parameter. Normal range: 90 to 140 mL/min (males), 80 to 125 mL/min (females)
Time Frame: Baseline and week 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 162 | 82
mL/min | 2.25 (15.53) | -0.93 (11.36)

21. Other Pre Specified Outcome: Creatine Kinase (CK) - Change From Baseline to Week 16
Description: Creatine Kinase is a standard clinical chemistry parameter. Normal range: 35 to 232 U/L (males), 26 to 145 U/L (females)
Time Frame: Baseline and week 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 162 | 82
U/L | 7.9 (64.9) | 5.6 (65.7)

22. Other Pre Specified Outcome: Erythrocytes (RBC) - Change From Baseline to Week 16
Description: Erythrocytes (red blood cells, RBC) is a standard clinical hematology parameter. Normal range: 4.6 to 5.8*10^12 cells/L (males), 4.1 to 5.2*10^12 cells/L (females)
Time Frame: Baseline and week 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: *10^12 cells/L
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 155 | 81
*10^12 cells/L | -0.14 (0.39) | 0.04 (0.31)

23. Other Pre Specified Outcome: Leukocytes (WBC) - Change From Baseline to Week 16
Description: Leukocytes (white blood cells, WBC) is a standard clinical hematology parameter. Normal range: 4.0 to 10.7*10^9 cells/L
Time Frame: Baseline and week 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: *10^9 cells/L
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 155 | 81
*10^9 cells/L | -0.55 (1.77) | 0.23 (1.69)

24. Other Pre Specified Outcome: Lymphocytes - Change From Baseline to Week 16
Description: Total lymphocytes is a standard clinical hematology parameter. Normal range: 1.0 to 4.0*10^9 cells/L
Time Frame: Baseline and week 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: *10^9 cells/L
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 154 | 79
*10^9 cells/L | -0.16 (0.48) | 0.00 (0.53)

25. Other Pre Specified Outcome: Neutrophils - Change From Baseline to Week 16
Description: Neutrophils is a standard clinical hematology parameter. Normal range: 1.6 to 7.4*10^9 cells/L
Time Frame: Baseline and week 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: *10^9 cells/L
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 154 | 79
*10^9 cells/L | -0.31 (1.55) | 0.26 (1.57)

26. Other Pre Specified Outcome: Hemoglobin - Change From Baseline to Week 16
Description: Hemoglobin is a standard clinical hematology parameter. Normal range: 13.5 to 17.5 g/dL (males), 12.0 to 16.0 g/dL (females)
Time Frame: Baseline and week 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 155 | 81
g/dL | -0.69 (1.17) | 0.02 (0.88)

27. Other Pre Specified Outcome: Hematocrit - Change From Baseline to Week 16
Description: Hematocrit is a standard clinical hematology parameter. Normal range: 40 to 52% (males), 36 to 46% (females)
Time Frame: Baseline and week 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Volume percentage of red blood cells
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 155 | 81
Volume percentage of red blood cells | -2.0 (4.1) | 0.5 (3.5)

28. Other Pre Specified Outcome: Potassium - Change From Baseline to Week 16
Description: Potassium is a standard clinical chemistry parameter. Normal range: 3.5 to 5.3 mmol/L
Time Frame: Baseline and week 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 161 | 82
mmol/L | -0.08 (0.48) | -0.02 (0.56)

29. Other Pre Specified Outcome: Urate - Change From Baseline to Week 16
Description: Urate is a standard clinical chemistry parameter. Normal range: 4.0 to 8.5 mg/dL (males, 16-59 years), 3.4 to 8.7 mg/dL (males, >60 years) 2.5 to 7.5 mg/dL (females)
Time Frame: Baseline and week 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 162 | 82
mg/dL | -0.405 (1.415) | 0.209 (1.577)

30. Other Pre Specified Outcome: Urea (BUN) - Change From Baseline to Week 16
Description: Urea (blood urea nitrogen, BUN) is a standard clinical chemistry parameter. Normal range: 4 to 25 mg/dL
Time Frame: Baseline and week 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 162 | 82
mg/dL | -0.60 (15.26) | 0.99 (13.62)

31. Other Pre Specified Outcome: Cystatin C - Change From Baseline to Week 16
Description: Cystatin C is a biomarker. Normal range: 0.53 to 1.01 ng/mL
Time Frame: Baseline and week 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 139 | 66
ng/ml | 16.1 (241.1) | 62.9 (198.0)

32. Other Pre Specified Outcome: Triacylglycerol Lipase - Change From Baseline to Week 16
Description: Triacylglycerol lipase is a standard clinical chemistry parameter. Normal range: 7 to 60 U/L
Time Frame: Baseline and week 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 162 | 82
U/L | -4.2 (12.9) | 0.1 (17.5)

33. Other Pre Specified Outcome: Arterial Partial Pressure of Carbon Dioxide (PaCO2) - Change From Baseline to Week 16
Description: Arterial partial pressure of carbon dioxide (PaCO2) is performed as part of the capillary or arterial blood gas analysis. If possible, no supplementary oxygen was given during the resting period and while blood samples were drawn.
Time Frame: Baseline and week 16
Population: Safety (SAF) - a randomized participant was valid for safety analyses if at least one dose of study medication was administered. Only participants with a baseline and at least one measurement on treatment (or up to two days after stopping treatment) were included in the analysis of blood gas parameters.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 151 | 80
mmHg | 0.34 (4.05) | 0.56 (4.52)

34. Other Pre Specified Outcome: Arterial Partial Oxygen Pressure (PaO2) - Change From Baseline to Week 16
Description: Arterial partial pressure of oxygen (PaO2) is performed as part of the capillary or arterial blood gas analysis. If possible, no supplementary oxygen was given during the resting period and while blood samples were drawn.
Time Frame: Baseline and week 16
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 151 | 80
mmHg | -3.01 (14.71) | -4.95 (12.05)

35. Other Pre Specified Outcome: Oxygen Saturation (SaO2) - Change From Baseline to Week 16
Description: Oxygen saturation (SaO2) is measured as part of the capillary or arterial blood gas analysis. Normal blood oxygen saturation is considered 95-100 percent. If possible, no supplementary oxygen was given during the resting period and while blood samples were drawn.
Time Frame: Baseline and week 16
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: Percentage of oxygen saturation
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 151 | 79
Percentage of oxygen saturation | -1.5 (4.4) | -3.1 (8.0)

36. Other Pre Specified Outcome: Mean PR Duration (PRmean) - Change From Baseline to Week 16
Description: PR duration was evaluated as part of the 12-lead electrocardiogram. electrocardiograms (ECGs) were recorded after the participant had been at rest for 15 minutes in a supine position.
Time Frame: Baseline and week 16
Population: Safety (SAF) - a randomized participant was valid for safety analyses if at least one dose of study medication was administered. Only participants with a baseline and at least one measurement on treatment (or up to two days after stopping treatment) were included in the analysis of ECG parameters.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 162 | 78
ms | -0.32 (14.21) | 0.87 (11.16)

37. Other Pre Specified Outcome: Mean QRS Duration (QRSmean) - Change From Baseline to Week 16
Description: QRS duration was evaluated as part of the 12-lead electrocardiogram. ECGs were recorded after the participant had been at rest for 15 minutes in a supine position.
Time Frame: Baseline and week 16
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 165 | 80
ms | -0.19 (4.49) | -0.05 (4.30)

38. Other Pre Specified Outcome: Mean QT Duration (QTmean) - Change From Baseline to Week 16
Description: QT duration was evaluated as part of the 12-lead electrocardiogram. ECGs were recorded after the participant had been at rest for 15 minutes in a supine position.
Time Frame: Baseline and week 16
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 123 | 53
ms | 1.19 (24.89) | -2.00 (25.56)

39. Other Pre Specified Outcome: Mean QTcB Duration (Bazett's Correction Formula, QTcB) - Change From Baseline to Week 16
Description: Bazett-corrected QTcB duration was evaluated as part of the 12-lead electrocardiogram. ECGs were recorded after the participant had been at rest for 15 minutes in a supine position.
Time Frame: Baseline and week 16
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 123 | 53
ms | -4.30 (14.44) | -0.51 (15.58)

40. Other Pre Specified Outcome: Mean QTcF Duration (Fridericia's Correction Formula, QTcF) - Change From Baseline to Week 16
Description: Fridericia-corrected QTcF duration was evaluated as part of the 12-lead electrocardiogram. ECGs were recorded after the participant had been at rest for 15 minutes in a supine position.
Time Frame: Baseline and week 16
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 123 | 53
ms | -2.34 (13.71) | -1.02 (13.29)

41. Other Pre Specified Outcome: Mean RR Duration (RRmean) - Change From Baseline to Week 16
Description: RR duration was evaluated as part of the 12-lead electrocardiogram. ECGs were recorded after the participant had been at rest for 15 minutes in a supine position.
Time Frame: Baseline and week 16
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 166 | 81
ms | 3.89 (132.02) | -14.00 (131.93)

42. Other Pre Specified Outcome: Mean Ventricular Rate (VRmean) - Change From Baseline to Week 16
Description: Ventricular rate was evaluated as part of the 12-lead electrocardiogram. ECGs were recorded after the participant had been at rest for 15 minutes in a supine position
Time Frame: Baseline and week 16
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Number analyzed (Participants) | 166 | 81
beats per minute (bpm) | -0.70 (11.96) | 1.60 (11.68)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected after signing the informed consent until 2 days after end of study treatment over a period of approximately 30 days.
Arm/Group | Riociguat (Adempas, BAY63-2521)_individual Dose Titration | Placebo
Serious Adverse Events (participants affected / at risk) | 34/173 | 14/88
Other Adverse Events (participants affected / at risk) | 146/173 | 67/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Riociguat (Adempas, BAY63-2521)_individual Dose Titration (N=173) | Placebo (N=88)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 1
Atrial tachycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 2
Cardiac failure (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 6 | 3
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Chronic right ventricular failure (Cardiac disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Oedema due to cardiac disease (General disorders) | 1 | 0
Catheter site haemorrhage (General disorders) | 2 | 0
Bronchitis (Infections and infestations) | 1 | 1
Erysipelas (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Light chain analysis increased (Investigations) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope (Nervous system disorders) | 4 | 3
Bipolar I disorder (Psychiatric disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 2 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypotension (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Riociguat (Adempas, BAY63-2521)_individual Dose Titration (N=173) | Placebo (N=88)
Anaemia (Blood and lymphatic system disorders) | 5 | 1
Bradycardia (Cardiac disorders) | 1 | 2
Palpitations (Cardiac disorders) | 6 | 4
Right ventricular failure (Cardiac disorders) | 2 | 2
Ventricular extrasystoles (Cardiac disorders) | 0 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 4
Abdominal discomfort (Gastrointestinal disorders) | 6 | 2
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Abdominal pain upper (Gastrointestinal disorders) | 5 | 3
Constipation (Gastrointestinal disorders) | 10 | 1
Diarrhoea (Gastrointestinal disorders) | 17 | 4
Dry mouth (Gastrointestinal disorders) | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 31 | 7
Dysphagia (Gastrointestinal disorders) | 6 | 0
Gastritis (Gastrointestinal disorders) | 6 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 | 0
Nausea (Gastrointestinal disorders) | 19 | 7
Vomiting (Gastrointestinal disorders) | 17 | 3
Asthenia (General disorders) | 3 | 3
Chest discomfort (General disorders) | 5 | 1
Chest pain (General disorders) | 6 | 4
Fatigue (General disorders) | 5 | 4
Oedema (General disorders) | 6 | 2
Oedema peripheral (General disorders) | 27 | 18
Pyrexia (General disorders) | 2 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 2
Bronchitis (Infections and infestations) | 5 | 2
Influenza (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 26 | 8
Rhinitis (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 10 | 4
Urinary tract infection (Infections and infestations) | 7 | 2
Respiratory tract infection (Infections and infestations) | 4 | 1
Activated partial thromboplastin time prolonged (Investigations) | 8 | 2
Blood bilirubin increased (Investigations) | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 2 | 2
Blood creatinine increased (Investigations) | 3 | 5
Blood potassium increased (Investigations) | 0 | 2
Blood urea increased (Investigations) | 1 | 3
Creatinine renal clearance decreased (Investigations) | 1 | 3
Gamma-glutamyltransferase increased (Investigations) | 1 | 2
International normalised ratio increased (Investigations) | 10 | 4
Gout (Metabolism and nutrition disorders) | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 5
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Dizziness (Nervous system disorders) | 39 | 11
Headache (Nervous system disorders) | 43 | 12
Hypoaesthesia (Nervous system disorders) | 4 | 1
Paraesthesia (Nervous system disorders) | 3 | 3
Tremor (Nervous system disorders) | 2 | 2
Restless legs syndrome (Nervous system disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 4 | 6
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 4
Flushing (Vascular disorders) | 7 | 2
Haematoma (Vascular disorders) | 2 | 2
Hypotension (Vascular disorders) | 15 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The embargo can be up to 6 months (equal to the 180 days), moreover if it is necessary the embargo period can be prolonged to expiry of priority year.